CLINICAL TRIAL: NCT06347874
Title: Comparison of Cryoablation of Intercostal Nerves to Erector Spinae Plane Catheters in Patients With Rib Fractures
Brief Title: Cryo Rib Fracture Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANES-2024-32820
Record Dates: First submitted 2024-03-25; First posted 2024-04-04 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Rib Fractures
MeSH Terms: conditions — Rib Fractures | interventions — Cryosurgery

STUDY DESIGN:
Intervention Model Description: This is a randomized prospective controlled trial. This will be single blinded trial. The individual doing the outcome assessments will be blinded. Randomization will be 1:1.
Who Masked: Outcomes Assessor
Masking Description: The individual doing the outcome assessments will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cryoablation (Experimental): Participants with rib fracture randomized to Cryoablation.
  Interventions: Drug: Cryoablation
- ESP catheter (Active Comparator): Participants with rib fracture randomized to ESP Catheter.
  Interventions: Drug: ESP Catheter

INTERVENTIONS:
Drug: Cryoablation — an injection of 1ml of 1% lidocaine per rib and ultrasound guided cryoablation of the intercostal nerves
  Arms: Cryoablation
Drug: ESP Catheter — an ultrasound guided erector spinae plane catheter with initial bolus of 30 mL of 0.25% bupivacaine followed by infusion of 0.2% ropivacaine at 10 mL per hour via programmed intermittent bolus.
  Arms: ESP catheter

SUMMARY:
The purpose of this study is to determine if patients with rib fractures who undergo cryoablation of the intercostal nerves have improved pain control 7 days from procedure when compared to those who have a ESP catheter.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are over 18 who have more than one ribs fractured.

Exclusion Criteria:

* Patients who have an exclusion to regional anesthesia.
* Patients who are pregnant via self-report or pregnancy test if they take one.
* Non-English speakers
* Patients who have cold urticaria
* Patients with bilateral fractures
* Patients currently intubated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2027-01-20 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
Maximum pain score on POD (Post Operative Day) 7 | 7 days post procedure
  Maximum pain score on POD (Post Operative Day) 7
Opioid Use | 30 days post procedure
  Opioid Use measured in MMEs
Functional Pain Scores | 30 days post procedure
  Functional Pain Scores on POD 0,1,2,3,4,5,6,7,and 30
Number of Patients using opioids at POD 30 | 30 days post procedure
  , Number of Patients using opioids at POD 30
Length of hospital stay | 30 days post procedure
  Length of hospital stay measured in days:hours:minutes
Number of patients returned home by POD 30 | 30 days post procedure
  Number of patients returned home by POD 30
time to first ambulation | 30 days post procedure
  time to first ambulation measured in days:hours:minutes
number of patients admitted to ICU | 30 days post procedure
  number of patients admitted to ICU
number of patients that required mechanical ventilation | 30 days post procedure
  number of patients that required mechanical ventilation
Pulmonary Function Testing. | 30 days post procedure
  Pulmonary Function Tests include spirometry. For patients with pulmonary function testing, the test results between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Hanson, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States